CLINICAL TRIAL: NCT01818661
Title: Longitudinal Multi-Modality Imaging in Progressive Apraxia of Speech
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Jennifer Whitwell, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-008988, 17-010087; R01DC012519-09 (NIH)
Record Dates: First submitted 2013-03-20; First posted 2013-03-26 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: PPA; Non-fluent Aphasia; Apraxia of Speech; Primary Progressive Non-fluent Aphasia; Primary Progressive Aphasia
Keywords: apraxia of speech; non-fluent aphasia; aphasia
MeSH Terms: conditions — Aphasia, Broca; Apraxias; Primary Progressive Nonfluent Aphasia; Aphasia, Primary Progressive; Aphasia | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tau positron emission tomography (PET) (Experimental): All subjects will receive Tau PET scan on approximately day 1 or day 2 of study to assess Tau burden in the brain.
  Interventions: Drug: AV-1451

INTERVENTIONS:
Drug: AV-1451 — This is used to assess Tau burden in the brain.

SUMMARY:
The study is designed to determine the relationship between structural and functional changes in the brain on imaging and progression of speech and language, neurological and neuropsychological features in patients with neurodegenerative apraxia of speech (AOS).

DETAILED DESCRIPTION:
Apraxia of Speech (AOS) is a disorder of speech motor planning and/or programming that affects the production of speech, characterized by slow speaking rate, abnormal prosody and distorted sound substitutions, additions, repetitions and prolongations, sometimes accompanied by groping, and trial and error articulatory movements. While AOS is commonly associated with vascular insults, it can be the predominant manifestation of neurodegenerative disease. Apraxia of speech can be the only manifestation of a neurodegenerative disorder. However, AOS very often co-occurs with aphasia, particularly a non-fluent aphasia (NFA) of the Broca's type; a language disorder, typically characterized by agrammatic, telegraphic or truncated spoken language, often accompanied by similar difficulties with written language. Patients with neurodegenerative AOS can have varying degrees of NFA, with the aphasia considered more severe than the AOS in some patients, but with the AOS dominant in others. It is extremely rare to have a patient that presents with NFA that does not also have AOS. Patients with isolated AOS can develop NFA over time, although in some patients the AOS remains isolated for as many as 8-10 years.

Patients with AOS can also develop dysarthria and other non-speech motor symptoms, such as extrapyramidal features, postural instability, extra ocular eye movement abnormalities and limb apraxia. Cognitive impairment can also develop, although is rarely an early feature of the disease. The syndrome is progressive with many patients eventually becoming mute.

Studies have shown that patients with neurodegenerative AOS can be pathologically heterogeneous, with some cases showing deposition of the microtubule associated protein tau, while others have deposition of the TAR DNA binding protein of 43kDa (TDP-43). Typical tau pathologies that are observed include corticobasal degeneration, progressive supranuclear palsy (PSP) and Pick's disease. Clinical features are currently unhelpful in predicting the underlying pathology in these cases, although there is a suggestion that cases with isolated or dominant AOS may be more likely to show tau pathology, particularly PSP.

This project will be the first to assess longitudinal multi-modality neuroimaging in subjects with neurodegenerative AOS. It will allow us to assess all aspects of disease progression in these subjects, including changes on neuroimaging, speech and language, neurological, and neuropsychological assessments, to get a complete picture of dysfunction and progression in these subjects. This project will also be the first to apply DTI and the recently developed technique of resting state fMRI to the study of this disease. These techniques are of great current interest to the field and provide, for the first time, a way of assessing underlying functional and structural connectivity across the brain. Both techniques provide important information about how disease progresses through the brain tissue and have huge potential to be important future biomarkers of many different neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* We will study subjects that fulfill clinical inclusion criteria for neurodegenerative AOS that have been seen and diagnosed at Mayo Clinic

Exclusion Criteria:

* Subjects with concurrent illnesses that could account for speech and language deficits, such as traumatic brain injury, strokes or developmental syndromes will be excluded.
* Women that are pregnant or post-partum and breast-feeding will be excluded. All women who can become pregnant must have a pregnancy test no more than 48 hours before the PET scan.
* Subjects will also be excluded if MRI is contraindicated (metal in head, cardiac pace maker, e.t.c.), if there is severe claustrophobia, if there are conditions that may confound brain imaging studies (e.g. structural abnormalities, including subdural hematoma or intracranial neoplasm), or if they are medically unstable or are on medications that might affect brain structure or metabolism,(e.g. chemotherapy).
* Subjects will also be excluded if they do not have an informant, or do not consent to research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
measurement of longitudinal change in neuroimaging and the correlation between change on serial imaging measures and concurrent change on longitudinal measures of clinical performance in neurodegenerative AOS with or without non-fluent aphasia (NFA) | approxiamtely 1-2 years after baseline imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Whitwell, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No